CLINICAL TRIAL: NCT05365932
Title: Prospective Longitudinal Study for the Evaluation of an Intra Auricular Device as a Treatment for Painful Temporo-Mandibular Disorders
Brief Title: Evaluation of an Intra Auricular Device as a Treatment for Painful Temporo-Mandibular Disorders
Acronym: IAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Valeria Donnarumma, Principal Investigator, Federico II University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 303/18
Record Dates: First submitted 2022-03-07; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Temporomandibular Disorder; Pain; Psychosocial Impairment; Myofascial Pain
Keywords: Pressure Pain Threshold; Intra auricular device
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TMD Pain group (Experimental): Arm included patients with TMD Pain intensity >3 on a VAS scale and with diagnosis of myofascial pain, either alone or in combination with arthralgia, headache attributable to TMD or with disc displacement with reduction. Participants had to be 18 years of age or older. All subjects had to wear the device for 6 months and it should not be used for more than 23 hours in a 24-hour period
  Interventions: Device: Intra auricular device (IAD)

INTERVENTIONS:
Device: Intra auricular device (IAD) — The Intra Auricular Device (IADs) are a pair of inconspicuous, custom fit auricular prosthetic devices.The ear inserts are manufactured using computer-aided design/computer-aided manufacturing (CAD/CAM) technology and are made from a liquid, photo-reactive acrylate (EShell 300), used in hearing aid shells and otoplastics for the last 10 years. They are designed to be placed into the outer third of the ear canals, and they have a small retraction post used to facilitate removal . A red or blue dot, respectively, indicates the right and the left side. The device do not interfere with hearing or speech

SUMMARY:
Background: An innovative, non-invasive, and reversible Intra Auricular Device (IAD) has recently been introduced to treat temporomandibular muscle and joint disorders.Aim: To evaluate the effects of the IAD on pain, psychosocial domain and Pressure Pain Threshold (PPT) of masticatory muscles in patients with TMD pain. Methods: Ten subjects with TMD pain and with pain intensity higher than 30 mm on a VAS scale were included in the study. Patients received the IAD and counselling. Assessments included questionnaires of the DC/TMD Axis II questionnaires (Characteristic Pain Index, Interference, Jaw Functional Limitation Scale, Patient Health Questionnaire 9, Patient Health Questionnaire 15, Generalized Anxiety Disorder scale, Oral Behavior Checklist and Oral Health Impact Profile-22, Axis I clinical examination and PPTs at baseline (T0), after one month (T1), three months (T2) and six months (T3) from the first use of the device. PPTs were measured at anterior temporalis muscles, masseter muscles and right thenar as a control site.The Shapiro-Wilk test was used for the normal distribution of data. The difference among the longitudinal timepoints for variable was analysed with ANOVA. Statistical significance was accepted at p < 0.05.

DETAILED DESCRIPTION:
The goal of ths study is to evaluate the effects of a new intra auricular device, the IAD, on pain, psychosocial domain and Pressure Pain Threshold (PPT) of facial muscles in patients with diagnosis of TMD pain according to the Diagnostic Criteria of Temporomandibular Disorders

ELIGIBILITY:
Inclusion Criteria:

* age >18
* TMD-pain diagnosed according to the DC/TMD (myalgia, myofascial pain, arthralgia, headache attributable to TMD)
* disc displacement with reduction

Exclusion Criteria:

* disc displacement without reduction
* intermittent locking
* degenerative TMJ disorder
* craniofacial anomaly
* history of prior TMJ
* orthognathic surgery
* recent (within the past six months) trauma to the face or jaw
* current, active orthodontic treatment
* severe mental health disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Change of Pain (evaluated with Characteristic pain intensity scale) | Six months from the first use of the device
  This questionnaire is a valid instrument assessing pain intensity, numbers of days with interference and pain-related disability in the last month. The characteristic pain intensity score, which ranges from 0-100, is calculated as the mean intensity ratings for reported current, worst, and average pain
Change of Pain evaluated with instrumental exam( Pain Pressure Threshold) | Six months from the first use of the device
  Pain Pressure Threshold were assessed by a single examiner at the anterior temporalis and masseter muscles (respectively TdxM; TsxM; MdxM; MsxM). An additional measurement was performed at the right thenar muscle (TenM) selected as a control muscular site.
Psychosocial domain positive change | Six months from the first use of the device
  Evaluation of psychosocial positive change through psychosocial questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Donnarumma Valeria, Afragola, Italy